CLINICAL TRIAL: NCT03995017
Title: A Phase I/II Trial of Rucaparib in Combination With Ramucirumab With or Without Nivolumab in Previously Treated Patients With Advanced Gastric and Esophageal Adenocarcinoma (RiME)
Brief Title: Rucaparib Plus Ramucirumab With or Without Nivolumab in Advanced Gastric and Esophageal Adenocarcinoma
Acronym: RiME
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Bristol-Myers Squibb (Industry); Clovis Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IIT-2018-RucaRamNivo
Record Dates: First submitted 2019-06-19; First posted 2019-06-21 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Esophagus Cancer, Adenocarcinoma; Stomach Cancer, Adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma Of Esophagus; Stomach Neoplasms; Adenocarcinoma | interventions — rucaparib; Ramucirumab; Nivolumab

STUDY DESIGN:
Intervention Model Description: Phase 1 - Safety Lead In - Enroll 6-9 molecularly unselected participants to determine the safety of the triplet combination of Rucaparib plus Ramucirumab and Nivolumab. One level dose de-escalation of Rucaparib will be planned based on dose limiting toxicity (DLT) signal of the first 6 participants run in phase.
  Phase 2 - Parallel - Enroll 52 participants (26 in each cohort), open label, two treatment cohorts design evaluating Rucaparib plus Ramucirumab with or without Nivolumab. 50 percent (%) of participants enrollment to each treatment cohort will represent molecularly unselected population and the remaining 50% will be selected based on integrated screening tumor Homologous Recombination Deficiency (HRD) gene panel. The primary objective is efficacy by measuring the Overall Response Rate (ORR).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Safety Lead In (Experimental): * Rucaparib 600 milligrams twice daily
  * Ramucirumab 8 milligrams per kilogram intravenous every 2 weeks
  * Nivolumab 480 milligrams intravenous every 4 weeks
  * Treatment will continue until disease progression, unacceptable toxicity or the patient desires to discontinue this therapy
  * One dose level decrease of Rucaparib will be planned if toxicity develops in the first 6 patients
  * 1 cycle= 28 days
  Interventions: Drug: Rucaparib; Drug: Ramucirumab; Drug: Nivolumab
- Cohort A (Experimental): * Rucaparib 600 milligrams twice daily
  * Ramucirumab 8 milligrams per kilogram intravenous every 2 weeks
  * Nivolumab 480 milligrams intravenous every 4 weeks
  * Treatment will continue until disease progression, unacceptable toxicity or the patient desires to discontinue this therapy
  * 1 cycle= 28 days
  Interventions: Drug: Rucaparib; Drug: Ramucirumab; Drug: Nivolumab
- Cohort B (Active Comparator): * Rucaparib 600 milligrams twice daily
  * Ramucirumab 8 milligrams per kilogram intravenous every 2 weeks
  * Treatment will continue until disease progression, unacceptable toxicity or the patient desires to discontinue this therapy
  * 1 cycle= 28 days
  Interventions: Drug: Rucaparib; Drug: Ramucirumab

INTERVENTIONS:
Drug: Rucaparib — Rucaparib tablet
  Other Names: Rubraca
Drug: Ramucirumab — Ramucirumab intravenous solution
  Other Names: Cyramza
Drug: Nivolumab — Nivolumab intravenous solution
  Other Names: Opdivo; Bristol- Meyers Squibb (BMS)-936558
  Arms: Cohort A; Safety Lead In

SUMMARY:
The study population is advanced gastric, gastroesophageal, and esophageal adenocarcinoma participants who have failed upfront standard of care chemotherapy. The goal is to demonstrate that Rucaparib plus Ramucirumab with or without Nivolumab has a higher response rate than what has been reported for Ramucirumab in previously treated patients. Trial will be a phase 1/2 trial. The Phase 1 portion will determine the recommended Phase 2 treatment dose for the combination of Rucaparib plus Ramucirumab and Nivolumab and enroll approximately 6-9 participants. The Phase 2 portion of the study will involve 52 participants allocated between two treatment groups comparing Rucaparib plus Ramucirumab with or without Nivolumab. The participants will be selected based on the results of a screening HRD gene panel.

ELIGIBILITY:
Inclusion Criteria:

* Half of the study population in phase 2 must have a deleterious tumor alteration in at least one protocol specified gene
* Gastric or gastroesophageal junction adenocarcinoma
* Advanced stage 4 or locally unresectable stage 3 disease
* Must have measurable disease
* Must consent to have a biopsy if archival tissue is not available or not enough for molecular testing
* Must show evidence of progression or intolerance to at least one previous standard of care systemic therapy (not more than 2 lines of prior therapy)
* Patients with human epidermal growth factor receptor 2 (HER2) positive disease must show progression on prior HER2 targeted therapy
* Toxicities related to prior treatment should be recovered to baseline or less than grade 2 according to CTCAE
* Adequate organ and marrow function
* Absence of active autoimmune disease that has required systemic treatment in the past 2 years
* Absence of conditions requiring systemic treatment with either corticosteroids or other immunosuppressive medications within 14 days of study drug administration. 10mg or less of prednisone or equivalent is acceptable
* Evidence of post-menopausal status or negative serum pregnancy test for female pre-menopausal patients
* Women of child-bearing potential and men with partners of child-bearing potential must agree to practice sexual abstinence, or to use two forms of adequate contraception prior to study entry, for the duration of study participation, and for 6 months following completion of therapy
* Men of child-bearing potential must not father a child or donate sperm while on this study and for 7 months after their last study treatment

Exclusion Criteria:

* Prior treatment with a programmed cell death protein 1 (PD1) or programmed death- ligand 1 (PD-L1) inhibitors
* Prior treatment with poly-(ADP-Ribose)polymerase (PARP)
* Patients with microsatellite instability (MSI) high or mismatch repair (MMR) deficient tumors
* Abdominal fistula, GI perforation, bowel obstruction, or intra-abdominal abscess within 6 months before first dose
* Evidence of active peptic ulcer disease, inflammatory bowel disease, diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, acute pancreatitis, acute obstruction of the pancreatic duct or common bile duct, or gastric outlet obstruction
* Inability to swallow tablets
* Uncontrollable ascites or pleural effusion
* Cavitating pulmonary lesion(s) or known endotracheal or endobronchial disease manifestation
* Clinically significant hematuria, hematemesis, or hemoptysis, or other history of significant bleeding within 12 weeks
* Lesions invading any major blood vessels
* Receipt of the last dose of anticancer therapy less than 28 days prior to the first dose of study drug
* Major surgery within 8 weeks before first dose of study treatment
* History of allogenic organ transplantation
* Active infection including tuberculosis, hepatitis B, hepatitis C, or human immunodeficiency virus. Patients with a past or resolved hepatitis B virus (HBV) infection are eligible. Patients positive for hepatitis C antibody are eligible only if polymerase chain reaction is negative for hepatitis C virus (HCV) RNA
* Receipt of live attenuated vaccine within 30 days prior to the first dose of study drug
* Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, or serious chronic gastrointestinal conditions
* Uncontrolled hypertension defined as sustained blood pressure (BP) > 150 mm Hg systolic or > 100 mm Hg diastolic despite optimal antihypertensive treatment
* Prolonged baseline QT interval corrected for heart rate greater than 470 ms
* Brain metastases or spinal cord compression. Patients whose brain metastases have been treated may participate provided they show radiographic stability
* Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients
* Current or anticipated use of other investigational agents while participating in this study
* History of another primary malignancy except for:

  * Malignancy treated with curative intent and with no known active disease before the first dose of investigational product (IP) and of low potential risk for recurrence
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  * Adequately treated carcinoma in situ without evidence of disease
* Psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-01-09 (Actual); Primary Completion 2022-10-19 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Recommended Phase 2 Dose (RP2D) | Up to 28 days
  Defined as the highest dose studied for which the observed incidence of dose limiting toxicities (DLT) is less than 33%. DLTs will be measured per the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Overall Response Rate (ORR) | up to 12 months
  Defined as the proportion of participants with overall response to therapy. Overall response is defined as the best response recorded, (including Complete Response (CR) and Partial Response (PR)), from the start of the treatment until the end of treatment. ORR will be measured per the Modified Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria

SECONDARY OUTCOMES:
Number of participants with treatment related adverse events (TRAEs) | Up to 12 months
  Determining per CTCAE 5.0
Overall Benefit Rate (OBR) | Up to 12 months
  Defined as the proportion of participants with overall benefit to therapy. Overall benefit is defined as the best response recorded, (including complete Response (CR), Partial Response (PR), and Stable Disease (SD)), from the start of the treatment until the end of treatment. Determine overall benefit of therapy using modified RECIST version 1.1
Progression free survival (PFS) | Up to 12 months
  Reported as the proportion of participants that achieve PFS. PFS is defined as the time from the start of treatment until the first documentation of disease progression or death due to any cause, whichever occurs first. Measured per modified RECIST version 1.1
Overall survival (OS) | Up to 12 months
  Defined as the time from the start of treatment until death due to any cause, reported as the mean of all participants' OS. Measured per the medical record.

CONTACTS AND LOCATIONS:
Overall Officials: Anwaar Saeed, MD, Principal Investigator — Kansas University Cancer Center
Locations (8):
- United States (8):
  - University of Chicago Medical Center, Chicago, Illinois
  - KU Cancer Center, Fairway, Kansas
  - University of Kansas Cancer Center - CRC, Fairway, Kansas
  - University of Kansas Cancer Center - West, Kansas City, Kansas
  - The University of Kansas Cancer Center, Westwood Campus, Kansas City, Kansas
  - University of Kansas Cancer Center - Overland Park, Overland Park, Kansas
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri

IPD SHARING:
Plan to Share IPD: No